CLINICAL TRIAL: NCT03965390
Title: Exploratory Study of Oral Therapeutic Education in Stimulated Parkinsonian Patients: Monitoring of Periodontal Status and Microbiota
Brief Title: Oral Therapeutic Education in Stimulated Parkinsonian Patients
Acronym: BUCCO-PARK
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: impossibility of continuing the study due to lack of medical staff
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 35RC18_8971_BUCCO-PARK
Record Dates: First submitted 2019-05-21; First posted 2019-05-29 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Parkinson Disease; Oral Infection
Keywords: oral microbiota; parkinson; brain stimulation surgery; oral therapeutic
MeSH Terms: conditions — Parkinson Disease | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Classical care pathway (No Intervention): Patients are following classical care pathway. Before brain surgery patients will be included after oral, medical and life quality evaluation.
  After randomization in the control group, patients will be evaluated at 6 and 12months after surgery, during classical follow up visits.
- Oral education (Experimental): Patients are following classical care pathway but combined at each visit with an oral education Before brain surgery patients will be included after oral, medical and life quality evaluation.
  After randomization in the experimental group, patients will be evaluated at 6 and 12 months after surgery, during classical follow up visits. At each timepoint an oral education will be realized in parallel.
  Interventions: Behavioral: Oral education

INTERVENTIONS:
Behavioral: Oral education — Oral therapeutic education aims to improve dietary practices, daily hygiene and care, in an approach adapted to the characteristics and consequences of Parkinson's disease. An oral prevention package will be given to patients.
  Initially, dentists expose various oral health problems commonly found in Parkinson's disease, in order to give patients the necessary information for the understanding Secondly, dentists dispenseront practical advice tailored to pathology, to maintain good oral health
  Arms: Oral education

SUMMARY:
The effect of periodontal disease on the general condition of patients remains today underestimated in Parkinson's disease. The BUCCO-PARK project aims to carry out an exploratory study of oral therapeutic education on the clinical evolution and fate of the microbiota of patients undergoing brain stimulation surgery. During the study, patients will follow the standard care pathway alone or combined with an oral therapeutic education. Biological samples will assess how the microbiota of these patients will be impacted. BUCCO-PARK aims to optimize the care of Parkinson's patients by integrating oral care.

DETAILED DESCRIPTION:
Patients included will be randomized in one of both defined groups : experimental group, in which patients will receive an oral education or control group, in which patient only follow the traditional care pathway.

Patients will be included in the trial before surgery after medical examination and life quality and oral environment evaluations.

Oral therapeutic education for patients randomized in experimental group will be performed at inclusion, and 6, and 12 months after surgery.

For all patients, an oral examination, an assessment of the quality of life and oral, fecal and blood samples will be carried out at inclusion, and 6 and 12 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with idiopathic Parkinson's disease for whom deep brain stimulation surgery (indifferent target) has been indicated for their Parkinson's disease
* affiliated to a system of social security;
* having at least 10 natural teeth (treated or not)
* having received oral and written information on the protocol and having signed a consent to participate in this research.

Exclusion Criteria:

* pregnant or lactating women;
* Persons of legal age subject to legal protection (safeguard of justice, guardianship, tutorship), persons deprived of their liberty;
* Patients who do not speak French (both written and spoken);
* Patients whose oral status is considered incompatible by the dental surgeon investigator with entry into the study (history of major maxillofacial surgery, presence of drugs that may cause gingival hypertrophy 2 or gingival bleeding 3).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-12-14 (Actual); Primary Completion 2023-05-19 (Actual); Study Completion 2023-05-19 (Actual)

PRIMARY OUTCOMES:
Parodontal disease progression after 12 months | 12 months
  Parodontal disease progression according to criteria defined by CDC/AAP 6 months after surgery

SECONDARY OUTCOMES:
Parodontal disease progression after 6 months | 6 months
  Parodontal disease progression according to criteria defined by CDC/AAP 6 months after surgery
Parodontal disease progression at inclusion | 1 month
  Parodontal disease progression according to criteria defined by CDC/AAP at inclusion
Caries index progression | 12 months
  Assessment of dental state using caries index (from 1 : low risk to 3) at inclusion and 6 and 12 months after surgery. Carious index measuring the number of decayed teeth, absent for decay and closed in permanent toothing.
Plaque index progression | 12 months
  Assessment of dental state using plaque index (from 0 : absence of microbial plaque to 3 : large amount of plaque in sulcus or pocket), at inclusion and 6 and 12 months after surgery. After all teeth are examined and scored, the index is calculated by dividing the number of plaque containing surfaces by the total number of available surfaces.
Gingival index progression | 12 months
  Assessment of dental state using gingival index at inclusion and 6, and 12 months after surgery. Gingivitis index is the number assigned to designate the degree of gingival inflammation. From 0 : Normal to 3 : Advanced gingivitis
Papillary bleeding index progression | 12 months
  Assessment of dental state using papillary bleeding index at inclusion and 6, and 12 months after surgery. The intensity of any bleeding is recorded as: Score 0 - no bleeding; to Score 4 - Profuse bleeding occurs after probing; blood flows immediately into the marginal sulcus.
Number of loss of attachment | 12 months
  Assessment of dental state using number of loss of attachment at inclusion and 6, and 12 months after surgery.
OHIP-14 score at inclusion | 1 month
  oral health impacts profile (OHIP-14) score at inclusion. Questionnaire with 14 items, each from 1 (no problem) to 5 (Locker et al. J Can Dent Assoc, 1993)
OHIP-14 score after 6 months | 6 months
  oral health impacts profile (OHIP-14) score 6 months after surgery. Questionnaire with 14 items, each from 1 (no problem) to 5 (Locker et al. J Can Dent Assoc, 1993)
OHIP-14 score after 12 months | 12 months
  oral health impacts profile (OHIP-14) score 12 months after surgery. Questionnaire with 14 items, each from 1 (no problem) to 5 (Locker et al. J Can Dent Assoc, 1993)
NMSS score at inclusion | 1 month
  Non Motor Symptoms Scale score at inclusion. Medical questionnaire with 30 items assessing symptoms progression. For each item, severity and frequency are assessed. Severity is assessed from 0 (no severity) to 3 and frequency from 1 (rare) to 4
NMSS score after 6 months | 6 months
  Non Motor Symptoms Scale score 6 months after surgery. Medical questionnaire with 30 items assessing symptoms progression. For each item, severity and frequency are assessed. Severity is assessed from 0 (no severity) to 3 and frequency from 1 (rare) to 4
NMSS score after 12 months | 12 months
  Non Motor Symptoms Scale score 12 months after surgery. Medical questionnaire with 30 items assessing symptoms progression. For each item, severity and frequency are assessed. Severity is assessed from 0 (no severity) to 3 and frequency from 1 (rare) to 4
alpha diversity of microbiota | 12 months
  alpha diversity is expressed as number of observed species of oral and intestinal microbiota at inclusion, and 6, and 12 months after surgery. Alpha diversity is defined by Whittaker (1972) as the species richness of a place. The higher the number, the higher the diversity.
beta diversity of microbiota | 12 months
  beta diversity is relative bacterial abundance at different levels in percent at inclusion, and 6, and 12 months after surgery. Beta diversity was defined by Whittaker (1972) as "the extent of species replacement or biotic change along environmental gradients. The higher the number, the higher the change is
Change in non-motor aspects of experiences of daily living (MDS-UPDRS I) | 12 months
  Change in non-motor aspects of experiences of daily living (MDS-UPDRS I) between the Baseline assessment and the assessment at 6, and 12 months' follow up The Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) is the standard validated tool for the assessment of patients with Parkinson's Disease (PD). This combined scale includes subsections collecting data regarding: nonmotor experiences of daily living (part I), their motor experiences of daily living (part II) an examination of the motor features of PD (part III), and motor complications arising from the use of dopamine replacement (part IV). The Part I include 13 items (6 semistructured interview items and 7 self-reported items) scored on a scale from 0 (normal) to 4 (severe). Higher scores reflect worse condition.
Change in motor aspects of experiences of daily in "on" and "off" medication (MDS-UPDRS II) | 12 months
  Change in motor aspects of experiences of daily in "on" and "off" medication (MDS-UPDRS II) between the Baseline assessment and the assessment at 6, and 12 months' follow up The Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) is the standard validated tool for the assessment of patients with Parkinson's Disease (PD). This combined scale includes subsections collecting data regarding: nonmotor experiences of daily living (part I), their motor experiences of daily living (part II) an examination of the motor features of PD (part III), and motor complications arising from the use of dopamine replacement (part IV). The Part II include 13 self-reported items) scored on a scale from 0 (normal) to 4 (severe). Higher scores reflect worse condition.
Change in motor examination during "on" periods (MDS-UPDRS III) | 12 months
  Change in motor examination during "on" periods (MDS-UPDRS III) between the Baseline assessment and the assessment at 6, and 12 months' follow up The Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) is the standard validated tool for the assessment of patients with Parkinson's Disease (PD). This combined scale includes subsections collecting data regarding: nonmotor experiences of daily living (part I), their motor experiences of daily living (part II) an examination of the motor features of PD (part III), and motor complications arising from the use of dopamine replacement (part IV). The Part III include 18 items scored on a scale from 0 (normal) to 4 (severe). Higher scores reflect worse condition.
Change in motor complications with MDS-UPDRS IV | 12 months
  Change in motor complications with MDS-UPDRS IV between the Baseline assessment and the assessment at 6, and 12 months' follow up The Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) is the standard validated tool for the assessment of patients with Parkinson's Disease (PD). This combined scale includes subsections collecting data regarding: nonmotor experiences of daily living (part I), their motor experiences of daily living (part II) an examination of the motor features of PD (part III), and motor complications arising from the use of dopamine replacement (part IV). The Part IV include 6 items assessed in a semistructured interview, scored on a scale from 0 (normal) to 4 (severe). Higher scores reflect worse condition.
Motor symptom evaluation using Hoehn and Yahr score | 12 months
  Motor symptom evaluation using Hoehn and Yahr stade. Hoehn and Yahr score evaluation at inclusion and 6 and 12 months after surgery. Hoehn and Yahr ladder defines 6 stages, from 0 (no parkinson signs) to 6 (no more autonomy). Reference : Hoehn et al. Neurology 1967
Ferric markers determination | 12 months
  Determination of ferric markers using ferric blood test results. Blood tests will be realized at inclusion and 6 and 12 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Marc VERIN, Pr, Principal Investigator — Rennes University Hospital
Locations (1):
- CHU de Rennes, Rennes, France